CLINICAL TRIAL: NCT03183674
Title: Oxytocin in Individuals With Spectrum Autism Disorders
Brief Title: Oxytocin in Spectrum Autism Disorders
Acronym: OxytocinASD
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of Sao Paulo General Hospital (Other)
Responsible Party: Principal Investigator, Helena Paula Brentani, Prof. DRa, University of Sao Paulo General Hospital
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Other
Other Study IDs: 10922213.7.0000.0068-2
Record Dates: First submitted 2017-05-23; First posted 2017-06-12 (Actual); Last update posted 2019-10-28 (Actual); Status verified 2019-10

CONDITIONS: Autistic Disorder
MeSH Terms: conditions — Autistic Disorder | interventions — Oxytocin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- oxytocin spray (Experimental): oxytocin nose spray dose 0,4IU/kg, once unique dose
  Interventions: Drug: Oxytocin
- placebo (Placebo Comparator): saline nose spray, 0,9 %, once unique dose
  Interventions: Other: placebo

INTERVENTIONS:
Drug: Oxytocin — Single dose oxytocin 45 minutes before the test
  Other Names: syntocinon
  Arms: oxytocin spray
Other: placebo — saline solution 0,9% spray nasal
  Arms: placebo

SUMMARY:
Observe effects of oxytocin on individuals with autism spectrum disorder

DETAILED DESCRIPTION:
To observe the effects of oxytocin on individuals with autism spectrum disorder according to gender, in facial recognition and eye tracking tests. The investigators will apply the nepsy and eye tracking tests before and 45 minutes after the puff with oxytocin or placebo at the dose of 0.4 IU / kg / dose maximum of 24 IU. The next week the volunteer will return and will do the same procedure because whoever took the placebo would take oxytocin and vice versa. Is a randomized, double-blind, placebo-controlled clinical trial.

ELIGIBILITY:
Inclusion Criteria:Diagnosis of ASD by DSMV

* CARS> 30
* age between 3 and 16 years
* stable (3 months with medication maintained or without medication)

Exclusion Criteria:- pregnant women, infants and

* participation in another research project of pharmacological or behavioral intervention in progress
* Use of pituitary hormones, cortisol, androgens and estrogens.
* heart problems: recent AMI, heart failure.
* respiratory problems: pneumonia, respiratory failure, decompensated asthma, acute bronchitis.

Ages: 3 Years to 16 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 80 (Actual)
Dates: Start 2016-07-15 (Actual); Primary Completion 2017-07-20 (Actual); Study Completion 2018-05-15 (Actual)

PRIMARY OUTCOMES:
Eye tracking | on average of 1 year
  Eye tracking program

SECONDARY OUTCOMES:
Nepsy | on average of 1 year
  face recognize

CONTACTS AND LOCATIONS:
Overall Officials: Debora Zambori, Study Chair — Instituto de Psiquiatria
Locations (1):
- Instituto de Psiquiatria, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: Yes
The investigators intend to share research information, such as, harms and benefits
Supporting Information: Study Protocol
Time Frame: 6 months
Access Criteria: Clinicians and students